CLINICAL TRIAL: NCT00834184
Title: Phase I, Randomized, Double-blind, Placebo Controlled, Multiple-dose Evaluation of the Safety Tolerance and Pharmacokinetics of Nikkomycin Z in Healthy Subjects
Brief Title: Safety and PK of Nikkomycin Z in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: VFCE-2008-002
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Healthy
Keywords: nikkomycin Z; pharmacokinetics; toxicity
MeSH Terms: interventions — nikkomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Experimental): nikkomycin Z 250 mg BID versus placebo BID x 14 days
  Interventions: Drug: nikkomycin Z
- B (Experimental): nikkomycin Z 500 mg BID versus placebo BID x 14 days
  Interventions: Drug: nikkomycin Z
- C (Experimental): nikkomycin Z 750 mg BID versus placebo BID x 14 days
  Interventions: Drug: nikkomycin Z
- D (Experimental): nikkomycin Z 750 mg TID versus placebo TID x 14 days
  Interventions: Drug: nikkomycin Z

INTERVENTIONS:
Drug: nikkomycin Z — Multiple rising doses. Doses packaged on a unit dose basis in 250 mg capsules. Subjects take 1-3 capsules per dosing block for 14 days unless ADE or study withdrawal. Dose escalation unless a dose-limiting adverse effect is noted. Subjects assigned to BID dosing will receive 28 doses and subjects assigned to TID dosing will receive 42 doses.
  250 mg BID (n=6) vs Placebo capsule BID (n=2), 500 mg BID (n=6) vs Placebo capsule BID (n=2), 750 mg BID (n=6) vs Placebo capsule BID (n=2), 750 mg TID (n=6) vs Placebo capsule TID (n=2) At least 4 subjects complete lower dose before randomization includes next higher dose, thus there are 4 arms for active intervention and corresponding placebos.

SUMMARY:
The purpose of this study is to determine if nikkomycin Z is safe when administered at different dose levels for 14 days. The study will also determine blood levels and urinary excretion of nikkomycin Z in relation to dose administered. Healthy patients will be eligible to participate and will be allocated to receive nikkomycin Z (various doses) or a placebo.

DETAILED DESCRIPTION:
This protocol will serve as a Phase I, randomized, double-blind, placebo controlled, multiple-dose study to evaluate the safety, tolerance and pharmacokinetics of nikkomycin Z. Nikkomycin Z has previously been studied in a single dose protocol in healthy male subjects. This study is designed to run in parallel to protocol VFCE-2007-001 to provide additional data on safety and pharmacokinetics. The study will involve a total of 32 subjects (6 active/2 placebo per group) with a multiple, rising dose strategy.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years and <= 40 years
* Male or Female (if female, must have a negative pregnancy test and agrees to use an acceptable contraception method)
* Able to understand study and give written informed consent
* Be determined healthy based on a medical and laboratory evaluation

Exclusion Criteria:

* Patients under the age of 18 years or over 40 years
* Inability to comprehend study and provide written informed consent
* Inability to comply with the study requirements
* History of or current evidence of major organ disease including:
* Renal disease - serum creatinine > 1.5 mg/dL, significant hematuria or proteinuria, known structural abnormality or chronic kidney disease
* Hepatic disease - active viral hepatitis, history of hepatitis B or hepatitis C, bilirubin > 2.0, ALT or AST above normal upper limit for laboratory, alcoholic liver disease, other chronic liver disease
* CNS disease or cognitive dysfunction - any past history of epilepsy, CNS infections, stroke, CNS bleed, severe headaches, major psychiatric illness, or current mental status changes
* Lung disease - history of severe asthma, COPD, pulmonary tuberculosis, or other major lung disease
* Cardiac disease - history or current evidence of ischemic coronary artery disease, myocardial infarction, heart failure, significant arrhythmia
* Gastrointestinal disease - presence of inflammatory bowel disease, difficulty swallowing, or any gastrointestinal problem that would limit taking oral medications or that may compromise absorption of oral medications
* Cancer - History of hematologic malignancy or solid tumor excluding basal cell carcinoma limited to the skin within the past 5 years
* History of autoimmune or inflammatory disease such as rheumatoid arthritis and lupus
* Any other history or evidence of disease that in the opinion of the physician would increase the risk for the subject for clinical trial participation
* Immunocompromised state - solid organ transplant, cancer chemotherapy, BMT with graft versus host disease, immunosuppressive therapy, or HIV infection
* Recent weight loss of greater than 10%
* Regular use of prescription medications, over-the-counter medications, or dietary/herbal supplements within 14 days of day 1. Occasional use of acetaminophen or over-the-counter NSAID within the 14 day window may be allowed at the P.I.'s discretion
* Subjects who received another investigational drug within 30 days of enrollment

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Determine safety and tolerance of nikkomycin Z in healthy subjects following administration of multiple doses. | four weeks

SECONDARY OUTCOMES:
Evaluate the multiple dose pharmacokinetics of nikkomycin Z in healthy subjects | two weeks

CONTACTS AND LOCATIONS:
Overall Officials: David E Nix, Pharm D, Principal Investigator — University of Arizona
Locations (1):
- Clinical & Translational Research Center - University of Arizona, Tucson, Arizona, United States